CLINICAL TRIAL: NCT00247962
Title: A Randomized, Double-Blind Study Evaluating the Safety and Efficacy of Etanercept and Sulphasalazine in Subjects With Ankylosing Spondylitis
Brief Title: Study Evaluating Etanercept and Sulphasalazine in Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-402
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Results first posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept; Sulfasalazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: etanercept
- B (Active Comparator)
  Interventions: Drug: sulphasalazine (SSZ)

INTERVENTIONS:
Drug: etanercept — 50 mg
  Arms: A
Drug: sulphasalazine (SSZ) — Sulphasalazine: The target dose for SSZ is 1.5 g (3 tablets) twice daily orally. Subject start the oral TA at 0.5 g daily for the first week and increase by 0.5 g every week until a daily dose of 3 g. Is achieved by the start of study week 5 of the study.
  Arms: B

SUMMARY:
The purpose of this study is to compare the efficacy of etanercept and sulphasalazine in the treatment of Ankylosing Spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ankylosing spondylitis
* Active ankylosing spondylitis

Exclusion Criteria:

* Complete ankylosis of spine
* Previous treatment with etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2005-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Italy, descresg@wyeth.com; Trial Manager, Principal Investigator — For Hungary, WPBUMED@wyeth.com; Trial Manager, Principal Investigator — For Czech Republic, WPPGCLI@wyeth.com; Trial Manager, Principal Investigator — For Australia, medinfo@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Austria, WPVIMED@wyeth.com; Trial Manager, Principal Investigator — For Spain, infomed@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Denmark, medinfonord@wyeth.com; Trial Manager, Principal Investigator — For Finland, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For Sweden, MedInfoNord@wyeth.com; Trial Manager, Principal Investigator — For UK/Great Britian, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For Ireland, ukmedinfo@wyeth.com; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For China, medinfo@wyeth.com
Locations (79):
- Australia (2):
  - Heidelberg West, Victoria
  - Shenton Park, Western Australia
- Austria (3):
  - Innsbruck
  - Klagenfurt
  - Linz
- China (2):
  - Beijing
  - Shanghai
- Czechia (2):
  - Ostrava
  - Prague
- Denmark (4):
  - Frederiksberg
  - Kolding
  - Odense
  - Vejle
- Finland (3):
  - Helsinki
  - Kuopio
  - Tampere
- France (9):
  - Amiens
  - Bordeaux
  - Boulogne-Billancourt
  - Créteil
  - Marseille
  - Nantes
  - Orléans
  - Pierre MendÃ¨s
  - Toulouse
- Germany (11):
  - Berlin
  - Erlangen
  - Gommern
  - Hamburg
  - Herne
  - Heubnerweg
  - Hildesheim
  - München
  - Pirna
  - Ratingen
  - Wiesbaden
- Hungary (5):
  - Debrecen
  - Győr
  - Nyíregyháza
  - Pécs
  - Szeged
- Ireland (2):
  - Wilton, Cork
  - Dublin
- Italy (8):
  - Benevento
  - Bergamo
  - Florence
  - Monserrato
  - Potenza
  - Prato
  - Reggio Emilia
  - Roma
- Netherlands (5):
  - Amsterdam
  - Groningen
  - Leeuwarden
  - Maastricht
  - Nijmegen
- Poland (4):
  - Lodz
  - Ustron Zawodzie
  - Warsaw
  - Wroclaw
- Doha, Qatar
- Riyadh, Saudi Arabia
- Spain (7):
  - Granollers, Barcelona
  - Asturias
  - Barcelona
  - Córdoba
  - Madrid
  - Porto
  - Santa Cruz de Tenerife
- Sweden (2):
  - Ostra Kyrkogardsgatan
  - Solna
- United Kingdom (8):
  - Upton, Wirral
  - Basingstoke
  - Cambridge
  - Cannock
  - Glasgow
  - Liverpool
  - Newcastle upon Tyne
  - Upper Borough Walls

REFERENCES:
- [Derived] Baraliakos X, Szumski AE, Kwok KK, Vlahos B, Borlenghi CE. Long-term Etanercept Response for Patients with Radiographic Axial Spondyloarthritis Based on Achievement of Early, Intermediate, or Late Responses During Index Studies. Rheumatol Ther. 2024 Jun;11(3):583-597. doi: 10.1007/s40744-024-00656-3. Epub 2024 Mar 15. PMID 38488976
- [Derived] Baraliakos X, Szumski A, Koenig AS, Jones H. The role of C-reactive protein as a predictor of treatment response in patients with ankylosing spondylitis. Semin Arthritis Rheum. 2019 Jun;48(6):997-1004. doi: 10.1016/j.semarthrit.2018.10.019. Epub 2018 Nov 2. PMID 30473179
- [Derived] Braun J, Pavelka K, Ramos-Remus C, Dimic A, Vlahos B, Freundlich B, Koenig AS. Clinical efficacy of etanercept versus sulfasalazine in ankylosing spondylitis subjects with peripheral joint involvement. J Rheumatol. 2012 Apr;39(4):836-40. doi: 10.3899/jrheum.110885. Epub 2012 Feb 15. PMID 22337244
- [Derived] Braun J, van der Horst-Bruinsma IE, Huang F, Burgos-Vargas R, Vlahos B, Koenig AS, Freundlich B. Clinical efficacy and safety of etanercept versus sulfasalazine in patients with ankylosing spondylitis: a randomized, double-blind trial. Arthritis Rheum. 2011 Jun;63(6):1543-51. doi: 10.1002/art.30223. PMID 21630245

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited in multiple countries from December 2005 to September 2007.
Pre-assignment Details: Subjects were screened up to 4 weeks in a 2:1 randomization ratio.
Groups:
- Etanercept: etanercept 50 mg once weekly
- Sulphasalazine: Sulphasalazine (SSZ) titration up to 3 g daily
Period: Overall Study
Arm/Group | Etanercept | Sulphasalazine
Started | 379 | 187
Completed | 353 | 168
Not Completed | 26 | 19
Not completed — Adverse Event | 15 | 12
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lack of Efficacy | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Sulphasalazine | Total
Number analyzed (Participants) | 379 | 187 | 566
Age Continuous [Mean (Standard Deviation); unit: years] | 40.69 (11.69) | 40.90 (12.23) | 40.76 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 47 | 147
  Male | 279 | 140 | 419
Region of Enrollment [Number; unit: participants]
  Qatar | 7 | 3 | 10
  Switzerland | 2 | 1 | 3
  Finland | 11 | 3 | 14
  Spain | 12 | 7 | 19
  Ireland | 1 | 0 | 1
  Austria | 3 | 1 | 4
  Italy | 19 | 8 | 27
  United Kingdom | 38 | 19 | 57
  France | 4 | 1 | 5
  Czech Republic | 36 | 18 | 54
  Hungary | 27 | 15 | 42
  Poland | 30 | 15 | 45
  Australia | 5 | 2 | 7
  Denmark | 13 | 6 | 19
  Netherlands | 7 | 4 | 11
  Germany | 62 | 31 | 93
  China | 17 | 9 | 26
  Sweden | 4 | 2 | 6
  Greece | 4 | 3 | 7
  Serbia | 54 | 27 | 81
  Mexico | 11 | 6 | 17
  Colombia | 8 | 4 | 12
  Portugal | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Assessment in Ankylosing Spondylitis (ASAS 20)
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) participants ASAS = 4 domains: participant global assessment of disease activity, pain, function, inflammation. ASAS 20 = 20% improvement from baseline and an improvement ≥ 10 units on a 0-100 scale (0=no disease activity; 100=high disease activity) for ≥ 3 domains, and no worsening in remaining domain.
Time Frame: 16 weeks
Population: All randomized patients who received at least 1 dose of study drug and had at least 1 post-baseline efficacy evaluation. Last observation carried forward approach (LOCF) used for missing data imputations.
Measure: Number; unit: participants
Arm/Group | Etanercept | Sulphasalazine
Number analyzed (Participants) | 378 | 187
participants | 287 | 99
Statistical Analysis 1: Comparison: Etanercept vs Sulphasalazine; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.99

2. Secondary Outcome: Ankylosing Spondylitis Quality of Life (ASQoL) Total Score Change From Baseline
Description: ASQoL is a questionnaire to assess disease specific quality of life. It consists of 18 statements that are relevant to the physical and mental conditions for a patient with Ankylosing Spondylitis (AS). Each statement is answered by the patients as a "Yes" (scored as 1) or "No" (scored as 0). All item scores are summed to give a total score. Scores can range from 0 (good QoL) to 18 (poor QoL).
Time Frame: Baseline and 16 Weeks
Population: The analysis population was limited to subjects whose native language was English, Hungarian and Dutch.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Sulphasalazine
Number analyzed (Participants) | 76 | 34
units on a scale
  Baseline | 11.03 (4.60) | 11.32 (4.75)
  Week 16 | 6.21 (5.31) | 9.06 (5.68)
Statistical Analysis 1: Comparison: Etanercept vs Sulphasalazine; baseline; Test type: Superiority or Other; p = 0.719, ANCOVA
Statistical Analysis 2: Comparison: Etanercept vs Sulphasalazine; week 16; Test type: Superiority or Other; p = 0.010, ANCOVA

ADVERSE EVENTS:
Arm/Group | Etanercept | Sulphasalazine
Serious Adverse Events (participants affected / at risk) | 7 | 4
Other Adverse Events (participants affected / at risk) | 213 | 100
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Etanercept | Sulphasalazine
Abdominal Pain (General disorders) | 0/379 | 1/187
Accidental Injury (General disorders) | 0/379 | 1/187
Migraine (Vascular disorders) | 1/379 | 0/187
Supraventricular Tachycardia (Cardiac disorders) | 1/379 | 0/187
Colitis (Gastrointestinal disorders) | 1/379 | 0/187
Gastritis (Gastrointestinal disorders) | 0/379 | 1/187
Arthritis (Musculoskeletal and connective tissue disorders) | 1/379 | 0/187
Dizziness (Nervous system disorders) | 0/379 | 1/187
Hypesthesia (Nervous system disorders) | 1/379 | 0/187
Neuralgia (Nervous system disorders) | 1/379 | 0/187
Paresis (Nervous system disorders) | 1/379 | 0/187
Psychosis (Nervous system disorders) | 0/379 | 1/187
Ptosis (Nervous system disorders) | 1/379 | 0/187
Vertigo (Nervous system disorders) | 1/379 | 0/187
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Etanercept | Sulphasalazine
Headache (General disorders) | 29/379 | 21/187
Injection Site Reaction (General disorders) | 41/379 | 3/187
Cardiovascular (Vascular disorders) | 23/379 | 10/187
Nausea (Gastrointestinal disorders) | 25/379 | 18/187
Metabolic and Nutritional (Metabolism and nutrition disorders) | 24/379 | 5/187
Nervous (Nervous system disorders) | 24/379 | 19/187
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 31/379 | 17/187
Skin and appendages (Skin and subcutaneous tissue disorders) | 39/379 | 14/187
Special Senses (Eye disorders) | 25/379 | 13/187

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.